CLINICAL TRIAL: NCT06957795
Title: Investigation of the Preoperative Effectiveness of Intensive Pelvic Floor Muscle Training in Women With Urinary Incontinence: a Randomized Controlled Trial.
Brief Title: Preoperative Pelvic Floor Muscle Training in Female Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-184
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Women; Urinary Incontinence (UI); Pelvic Floor Muscle Training; Preoperative Period
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patients in the control group will receive only pelvic floor knowledge and awareness training. Brief training on the functions and anatomy of the pelvic floor muscles and the function of the exercises performed, and will be taught how to contract their pelvic floor muscles. In the 6th week, all patients will be called for a final check-up and all the evaluations re-made.
- Exercise group (Experimental): Exercise group first receive brief training on the functions and anatomy of the pelvic floor muscles and the function of the exercises performed, and will be taught how to contract their pelvic floor muscles. In addition to this training, patients in exercise group will be taught pelvic floor exercises targeting the fast (tap) and slow twitch fibers (elevator) of the pelvic floor. The patients will do the exercises as a home program, and they will be called for an interim check-up in the 2nd week to check whether they are doing the exercises correctly and ensure their progress in the program. In the 6th week, all patients will be called for a final check-up and all the evaluations re-made.
  Interventions: Other: Intensive Pelvic Floor Exercise Program

INTERVENTIONS:
Other: Intensive Pelvic Floor Exercise Program — Intensive pelvic floor exercise program targeting the fast (tap) and slow twitch fibers (elevator) of the pelvic floor. The tap exercise will be performed by instructing the patient to quickly contract and release the pelvic floor muscles. For the elevator exercise, the patient will be asked to contract the pelvic floor muscles for 5 seconds and hold them for 5 seconds and then slowly relax them within 5 seconds. Patients will do the exercises as a home program. The exercise program will last for 6 weeks. One set of exercise will be counted as 10 taps and 10 elevator. In the first week, patients will be asked to do 5 sets of exercises per day and the number of sets will be increased by five for 6 weeks.
  Arms: Exercise group

SUMMARY:
Pelvic floor muscles (PFM) play a crucial role in supporting pelvic organs and maintaining continence. Weakness in these muscles can lead to dysfunctions such as pelvic organ prolapse, urinary incontinence (UI), and sexual or anorectal disorders. UI, defined as the involuntary loss of urine, is common globally and classified as stress, urge, or mixed incontinence. Stress urinary incontinence (SUI) - the most prevalent type among women - occurs during activities that increase intra-abdominal pressure. Risk factors include female sex, aging, obesity, smoking, chronic constipation, previous gynecological surgeries, and childbirth. Treatment options for SUI include conservative and surgical methods. Pelvic floor training (PFT), first described by Arnold Kegel in 1948, is a conservative approach that strengthens PFM and alleviates symptoms. Although surgery is often used for SUI, with over 200 procedures described, this study aims to evaluate the preoperative effectiveness of intensive PFT in women with SUI. It will assess changes in muscle function and symptoms before surgery, guiding pelvic rehabilitation strategies to potentially reduce surgical burden and improve outcomes.

DETAILED DESCRIPTION:
Pelvic floor muscles (PFM); is a muscle group that supports the pelvic organs like a hammock and has an important role in micturition and defecation. With the weakening of the PFM, dysfunctions such as pelvic organ prolapse (POP), chronic pelvic pain, anorectal dysfunction, sexual dysfunction and urinary incontinence can be observed. Urinary incontinence (UI), according to the definition of the International Continence Society (ICS), is the complaint of involuntary urine loss. UI can be seen in all ages and gender groups. UI affects people socially, physically and psychologically, as well as negatively affecting their quality of life. The prevalence of UI worldwide has been shown to be between 5.8% and 45.8%. It is reported that the prevalence of UI in Türkiye is between 26.3% and 71.5%. ICS examines urinary incontinence under 6 main headings, and the most common types are; stress, urgency and mixed type incontinence. Urinary incontinence characterized by a sudden, compelling desire to urinate is called urgency urinary incontinence (UUI); incontinence accompanied by increased abdominal pressure such as sneezing, coughing, laughing or lifting heavy objects is called stress urinary incontinence (SUI); and the occurrence of both symptoms together is called mixed type incontinence (MUI). Risk factors for incontinence include being a woman, smoking and having chronic constipation, advanced age, obesity, previous gynecological surgeries, pregnancy and childbirth. The most common type of urinary incontinence in women is SUI, known as involuntary urine loss during activities that increase intra-abdominal pressure such as coughing, laughing and lifting heavy objects. The treatment of SUI consists of conservative and surgical treatment options. The aim of surgical treatment is to correct the position of the urethra. Although surgical treatment is an effective method, it has some disadvantages such as the necessity of a long recovery period, recurrence of incontinence in 10%-40% of those who undergo surgery due to SUI, an increase in UUI after surgery, and high cost. In addition, conservative methods have gained importance in the treatment of SUI in recent years due to reasons such as some women not wanting to take surgical risks or surgical treatment not being applicable due to other systemic diseases. The aim of conservative treatment is to increase cortical awareness and muscle strength by increasing the strength of the pelvic floor muscles (PFM). PFM strengthening is important for the support of the pelvic organs and increasing the effectiveness of sphincteric activity around the urethra. Conservative treatment includes PFM (Kegel) exercises, vaginal weighting, electrical stimulation, and biofeedback-assisted PFM exercises to increase PFM strength and endurance. PFM exercises are included in all guidelines as the first choice treatment in the treatment of SUI (Evidence Level A). Biofeedback and PFM exercises are especially recommended for the treatment of SUI and MUI because they have no potential for side effects and are low-cost.

PFM exercises were first described by Arnold Kegel in 1948. Studies in the literature have shown that PFM exercises provide adequate muscle tone and function in female patients with SUI and regress SUI symptoms. The number of contractions in PFM exercises applied in studies varies from 8 to 12 contractions 3 times a day to 20 contractions 4 times a day or 200 contractions per day. However, there is no consensus on the most successful PFM exercise protocol.

Surgical treatment is often used for the treatment of urinary incontinence. More than 200 surgical methods have been described in the surgical treatment of SUI. Almost all of these surgical methods consist of approaches that support the midurethral and bladder neck and both vaginal and abdominal techniques. Strategies to improve outcomes in women undergoing surgery for urinary incontinence and/or pelvic organ prolapse would be beneficial to both patients and healthcare providers, as costs and burden of disease would be reduced. Preoperative and postoperative physiotherapy interventions can improve physical outcomes and quality of life in women undergoing/having surgery for urinary incontinence. In other areas, such as orthopedic surgery, physiotherapy is often initiated as a rehabilitation treatment before surgery and resumed as soon as possible after surgery to prevent loss of function. It has been reported in the literature that damage to the pubococcygeus muscle during prolapse surgery may contribute to the development of postoperative stress incontinence in previously continent patients, and that this can be prevented with physiotherapy. Despite this, there is no consensus in the urogynecology community on the role of physiotherapy in patients who are planned to undergo surgical correction of prolapse and/or incontinence. To our knowledge, there is no study on the effectiveness of intensive PFM exercises applied in the preoperative period in women with SUI and planned surgery. The aim of this study is to examine the effect of an intensive PFM exercise program applied in the preoperative period to women with SUI who are planned to undergo surgery on the level of pelvic floor knowledge, pelvic floor muscle function, pelvic floor symptoms and the rate of undergoing surgery. This study will reveal the changes in muscle function and symptoms caused by PFM exercises applied in the preoperative period in women who are planned to undergo SUI surgery. In addition, the effect of this exercise protocol applied in the preoperative period on the surgical needs of women will also be determined and will guide the planning of pelvic physiotherapy and rehabilitation programs to be applied before gynecological surgery to reduce surgical burden.

The type of study is a prospective, randomized controlled study. Our study will be conducted on women with complaints of SUI and SUI-dominant MUI and planned for surgery. Women who applied to the Department of Obstetrics and Gynecology, Gülhane Education and Research Hospital with complaints of urinary incontinence and were diagnosed with SUI or SUI-dominant MUI by their obstetrician-gynecologist will be included in the study. Patients will be divided into two groups by block randomization method in order to participate in the pelvic floor exercise program. A semi-structured assessment form will be used to record demographic data. Patients' age (years), height (cm), body weight (kg), education level, and marital status will be recorded. In addition, patients occupation, main complaint, duration of complaint, previous surgeries, and family history will be questioned, and their medications, obstetric history (number of pregnancies, number of births, type of birth), smoking, chronic cough, and constipation will be questioned. Pelvic floor evaluations of patients will be performed in a sterile and quiet room. Pelvic floor knowledge level will be determined with the Pelvic Floor Health Knowledge Test, pelvic floor muscle function will be determined manually according to the Modified Oxford Scale and perineometric measurement using a vaginal probe. In addition, pelvic floor symptoms and the level of discomfort felt from these symptoms will be evaluated with the Global Pelvic Floor Disorder Questionnaire and urinary incontinence severity will be evaluated with the Incontinence Severity Index. Whether or not women underwent surgery after treatment will be checked and recorded from the physician's record system. In order to follow the patients' compliance with the exercise, each patient will be given an exercise diary and asked to fill it out. The pre- and post-treatment evaluation data obtained will be determined by making intergroup and intragroup comparisons with the appropriate statistical method.

Individuals who agree to participate in the study will be included in the study after signing the written consent form. The intervention group of the women will be determined in a computer environment using the block randomization method. The sample size of this study was calculated as a total of 60 people, 30 in each group, using the G*Power 3.1 program, according to similar studies in the literature, with 80% power and a type 1 error level of 0.05.

ELIGIBILITY:
Inclusion criteria for the study:

* Being a woman between the ages of 18-65
* Being diagnosed with SUI or SUI-predominant mixed type urinary incontinence by an obstetrician-gynecologist
* Having active pelvic floor muscle contraction
* No genital anatomical abnormality
* Being able to understand and follow verbal and written instructions
* The patient was referred to physiotherapy at least 6 weeks before the planned surgery date
* Patients performed 75% or more of the given exercises (categorized as adequate compliance)

Exclusion criteria for the study:

* Not volunteering to participate
* Being pregnant
* Having had previous pelvic floor surgery
* Having received previous pelvic floor physiotherapy
* Having a vaginal or urinary infection
* Being unable to tolerate pelvic floor muscle function measurement
* Having a neuromuscular or neurological disease that may affect muscle function

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Symptoms | Before treatment, after treatment (end of 6 weeks)
  The severity of the symptoms of the patients will be evaluated with the Global Pelvic Floor Disorder Questionnaire measures the symptoms of stress urinary incontinence, urge urinary incontinence, frequent and sudden urination, difficulty urinating, pelvic organ prolapse, fecal incontinence, dyspareunia and obstructive defecation due to pelvic floor dysfunction and the discomfort felt from these symptoms. The scale consists of a total of 9 questions. The subjects were rated as "yes" or "no" (0) according to whether they had the complaint or not, and if they answered yes, they were rated as "not at all" (1), "very little" (2), "a little" (3), "quite a bit" (4), "a lot" (5). Each question was given a score between 1 and 5. The scoring system gives the same weight to each question. The total score is between 0 and 45. In order to score between 0 and 100, the average of the total score was taken and multiplied by 20. A high score indicates that the complaint is severe.
Change in Pelvic Floor Muscle Function | Before treatment, after treatment (end of 6 weeks)
  Change in pelvic floor muscle function of the patients will be evaluated with Modified Oxford grading system, a method frequently used in the clinic, will be used to evaluate pelvic floor muscle strength. While the patient is in the lithotomy position, two fingers will be placed in the vagina by an experienced physiotherapist. During this time, the patient will be asked to squeeze the muscles around the vagina as hard as she can. Contraction degree According to the Modified Oxford Scale, 0: No contraction, 1: Minimal contraction (able to hold the fingers for less than 1 second), 2: Weak contraction (no elevation of the fingers and able to hold for 1-3 seconds), 3: Moderate contraction (fingers are elevated to the posterior vaginal wall, can hold for 4-6 seconds), 4: Good contraction (Therapist's fingers are elevated to the posterior vaginal wall).
Change in Pelvic Floor Muscle Contraction | Before treatment, after treatment (end of 6 weeks)
  Pelvic floor muscle strength and endurance will be assessed using vaginal perineometry (Peritron™; Cardio-Design, Australia). The patient will lie on her back with hips and knees flexed and feet on the bed. She will be instructed not to hold her breath, not to contract abdominal, hip, or leg muscles, not to strain outward, take a deep breath, or move her pelvis during contraction. After confirming proper technique, the perineometer sensor will be inserted vaginally. The patient will be asked to contract and sustain the contraction of her pelvic floor muscles as long as possible, then relax without bearing down. Resting pressure, peak contraction pressure, and contraction duration (in seconds) will be recorded. Each measurement will be repeated three times, and average values will be used for analysis.
Change in Incontinence Severity | Before treatment, after treatment (end of 6 weeks)
  The incontinence severity assessment of the participants was made with the Incontinence Severity Index. Scale consists of two sub-items. These are determined as 'How often do you leak urine?', 'How much urine do you leak each time?' The score is obtained by multiplying the numbers of the questions in both items. The score will be determined by grouping them as 1-2 mild, 3-6 moderate, 8-9 severe, and 12 very severe.
Change in Pelvic Floor Health Knowledge | Before treatment, after treatment (end of 6 weeks)
  Pelvic Floor Health Knowledge Test was developed in Turkish and its reliability and validity have been demonstrated. Pelvic Floor Health Knowledge Test is given as "No" and "I don't know". Each correct answer is given "1" point, while incorrectly answered or unknown items are given "0" points, and as the score increases, it is an indication that the level of knowledge is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Education and Research Hospital, Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)